CLINICAL TRIAL: NCT04087694
Title: Comparative Study Between Microdecompression and Open Decompression With Posterior Stabilization for Symptomatic Lumbar Spine Stenosis
Brief Title: Microdecompression Versus Open Laminectomy and Posterior Stabilization for Multilevel Lumbar Spine Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Sherwan Ahmed Ali Hamawandi, Assistant professor of orthopedic surgery, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMU/SHERWAN
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Microdecompression; laminectomy; pain; stenosis
MeSH Terms: conditions — Spinal Stenosis; Pain; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open (Other): Open laminectomy and posterior stabilization with pedicle screws for symptomatic lumbar spine stenosis
  Interventions: Procedure: Microdecompression
- Microscope (Other): Microscopically done decompression of lumbar spine stenosis who are symptomatic
  Interventions: Procedure: Microdecompression

INTERVENTIONS:
Procedure: Microdecompression — comparative surgical treatment
  Other Names: Open decompression with posterior fixation

SUMMARY:
This study compare the results of 2 methods in surgical treatment of Lumbar spine stenosis.These are microdecompresssion and open decompression with posterior stabilization. 100 patients are involved in this study who divided in 2 groups.Each group was treated with one method and follow up done which showed both method are effective with better results in those patients treated with microdecomppression.

DETAILED DESCRIPTION:
This randomized controlled study was conducted between January 2016 and October 2018. One hundred patients were involved in this study. All these patients were suffered from radicular leg pain with MRI features of multilevel lumbar spinal stenosis and were treated by conservative treatment of medical treatment and physiotherapy without benefit for (6) months. Those patients were divided into two groups; Group A, (50) Microdecompression, and Group B, (50) patients who were treated by open wide laminectomy and posterior stabilization. Both groups of patients were followed up with ODI (Oswestry disability index) and VAS (Visual analogue score) for the back and leg pain for one year.

Results: The results showed that both groups got significant improvement regarding Oswestry disability index. Regarding back pain, there was a significant improvement in both groups with better results in-group A due minimal tissues injury as the advantage of minimal invasive technique. In both groups, there were marked improvement of radicular leg pain postoperatively.

Conclusions: Both Microdecompression and wide open laminectomy with posterior stabilization were effective in treatment of multilevel lumbar spinal stenosis with superior results of Microdecompression regarding less back pain postoperatively with less blood loss and soft tissue dissection.

ELIGIBILITY:
Inclusion Criteria:

* patients were suffered from back pain of different degrees with spinal claudication

Exclusion Criteria:

* Smoking
* Diabetic patients,
* Previous spinal surgery,
* any neuromuscular disorder like poliomyelitis, and
* vertebral instability proved by Dynamic plain radiographs

Ages: 41 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01-03 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Oswestry disability index | It was measured at 12 months after operation
  For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. If all 10 sections are completed the score is calculated as follows:
  Example: 16 (total scored) 50 (total possible score) x 100 = 32% If one section is missed or not applicable the score is calculated: 16 (total scored) 45 (total possible score) x 100 = 35.5% Minimum detectable change (90% confidence): 10% points (change of less than this may be attributable to error in the measurement)
Visual analoge score | It was measured at 12 months after operation
  This is in pain measurement ranging from 0 when no pain to 10 when there is severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Sherwan Hamawandi, Principal Investigator — Hawler medical university / college of medicine

IPD SHARING:
Plan to Share IPD: No
I want to share all my research with other researcher

REFERENCES:
- [Derived] Hamawandi SA, Sulaiman II, Al-Humairi AK. Microdecompression versus Open Laminectomy and Posterior Stabilization for Multilevel Lumbar Spine Stenosis: A Randomized Controlled Trial. Pain Res Manag. 2019 Nov 7;2019:7214129. doi: 10.1155/2019/7214129. eCollection 2019. PMID 31827656